CLINICAL TRIAL: NCT00221481
Title: An Evaluation of Divalproex vs. Olanzapine for Alcohol Abuse Relapse Prevention in Patients With Bipolar Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Mayo Clinic (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mark Frye, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 00-12-071-11A
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2009-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Alcohol
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Olanzapine

INTERVENTIONS:
Drug: divalproex or olanzapine

SUMMARY:
This study will evaluate how effective mood stabilizers are in the treatment of bipolar disorder with comorbid alcoholism

DETAILED DESCRIPTION:
Bipolar affective disorder is a medical illness with substantial morbidity and mortality. Further fueling the severity of this illness is the substantial co-occurrence with substance abuse that together poses an enormous public health problem.

This study will evaluate the efficacy of divaproex sodium (DVPX) vs. olanzapine (ZYP) vs. for alcohol relapse prevention and secondary mood stabilization. Bipolar patients who are actively drinking will be randomized to either Depakote ER ® (flexible dose schedule up to 2500 mg) or Zyprexa® (flexible dose schedule up to 20 mg). Adjunctive benzodiazepine will be utilized for the treatment of alcohol withdrawal and as an adjunct anxiolytic during the early titration of DVPX and ZYP. Patients who, after 2 weeks, have stabilized will continue in the prophylaxis study which will last up to 46 weeks. Flexible dose scheduling and adjunctive antidepressant treatment as clinically indicated will be done to maximize tolerability, treatment compliance, and mood stability.

The primary outcome measure will be alcohol abuse relapse which will be defined, a priori, as 5 drinks in a 24 hour period. Patients who have a relapse as such defined will be terminated from the study. Secondary alcohol outcome measures (i.e. number of drinking days, % drinking days per month, standard drinks per drinking occasion, craving) will be assessed through the time-line follow-back method. Secondary outcome measures of mood stabilization (major mood relapse and adjunctive medication) will be assessed by prospective life charting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* DSM-IV criteria for manic episode based on the SCID (Spitzer 1996)
* DSM-IV criteria for alcohol dependence or abuse based on the SCID. Meeting criteria for polysubstance dependence or abuse will not be exclusionary.
* Alcohol dependence/abuse confirmed by corroboration.
* Negative urine pregnancy test l

Exclusion Criteria:

* Inability to give informed consent
* Liver function tests greater than 3X the upper limit of normal
* History of adverse reaction to divalproex sodium or olanzapine
* History of seizure other than directly associated with prior alcohol withdrawal
* History of major head trauma with LOC > 5 minutes or skull fracture
* History of hypertension, neurologic illness
* Active hepatitis, hepatic encephalopathy, or history of pancreatitis
* Not practicing a reliable form of birth control

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frye, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Neuropsychiatric Institute, Los Angeles, California, United States